CLINICAL TRIAL: NCT00849472
Title: A Phase II Clinical Trial of Four Cycles of Doxorubicin and Cyclophosphamide Followed by Weekly Paclitaxel Given Concurrently With Pazopanib as Neoadjuvant Therapy Followed by Postoperative Pazopanib for Women With Locally Advanced Breast Cancer
Brief Title: Treatment With Pazopanib for Neoadjuvant Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110264; NSABP FB-6 (Other: National Surgical Adjuvant Breast and Bowel Project (NSABP))
Record Dates: First submitted 2009-02-12; First posted 2009-02-23 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2013-12

CONDITIONS: Neoplasms, Breast
Keywords: Neoadjuvant Breast Cancer; Pazopanib (GW786034); NSABP Foundation, Inc.; cyclophosphamide; Paclitaxel; Doxorubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — AC protocol; Paclitaxel; pazopanib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): Preoperative
  Cycles 1-4 Doxorubicin 60 mg/m2 IV over 15 minutes + Cyclophosphamide 600 mg/m2 IV over 30 minutes of Day 1 every 21 days
  followed by:
  Cycles 5-8 Paclitaxel 80 mg/m2 IV over 60 minutes (Days 1, 8, and 15) every 28 days in combination with pazopanib (800 mg) PO once daily (2 tablets taken at the same time each day either 1 hour before or 2 hours after a meal) Daily beginning on Day 1 of the first paclitaxel cycle Until 7 days before surgery
  Followed by Surgery
  Postoperative Pazopanib 800 mg PO once daily (2 tablets taken at the same time each day either 1 hour before or 2 hours after a meal) Daily beginning 4-6 weeks after surgery 6 months from first postoperative dose
  Interventions: Drug: doxorubicin + cyclophosphamide; Drug: paclitaxel + pazopanib; Procedure: surgery; Drug: pazopanib monotherapy

INTERVENTIONS:
Drug: doxorubicin + cyclophosphamide — 4 cycles of doxorubicin + cyclophosphamide followed by 4 cycles of paclitaxel + pazopanib.
Drug: paclitaxel + pazopanib — 4 cycles of paclitaxel + pazopanib
Procedure: surgery — neoadjuvant surgery for breast cancer
Drug: pazopanib monotherapy — 6 months of treatment with pazopanib monotherapy

SUMMARY:
The purpose of this study is to determine whether the treatment of a doxorubicin in combination with cyclophosphamide followed by a combination of pazopanib in combination with paclitaxel prior to surgery results in a pathological complete response in females with breast cancer.

DETAILED DESCRIPTION:
This is a phase II non-randomized, multi-center study aimed to evaluate the efficacy and safety of the combination of pazopanib and paclitaxel following treatment with cyclophosphamide and doxorubicin for the treatment of neoadjuvant breast cancer.

Patients will receive standard doses of AC every 21 days for 4 cycles. This will be followed by weekly paclitaxel 80 mg/m2 IV on Days 1, 8, and 15 every 28 days for 4 cycles given concurrently with pazopanib 800 mg PO daily starting with the first paclitaxel dose and continuing until 7 days before surgery. Clinical complete response rate will be determined by tumor assessments performed by palpation at two time points: following AC (before paclitaxel/pazopanib begins) and 2-4 weeks following the last dose of paclitaxel (before surgery). Following recovery from preoperative therapy, patients will undergo the clinically-indicated surgery. Pazopanib will resume 4-6 weeks after surgery and continue daily for 6 months of postoperative pazopanib therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and must have signed and dated an appropriate IRB-approved consent form that conforms to federal and institutional guidelines for the study treatment and submission of tumor and blood samples required for the FB-6 correlative science studies
* The ECOG performance status must be 0 or 1
* Patients must have the ability to swallow oral medication.
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or limited incisional biopsy.
* Patients must have ER analysis performed on the primary tumor prior to randomization. If ER analysis is negative, then PgR analysis must also be performed. (Patients are eligible with either hormone receptor-positive or hormone receptor-negative tumors.)
* Patients must have clinical stage IIIA, IIIB, or IIIC disease with a mass in the breast or axilla measuring at least 2.0 cm by physical exam, unless the patient has inflammatory breast cancer, in which case measurable disease by physical exam is not required.
* Adequate organ function
* LVEF assessment by 2-D echocardiogram or MUGA scan performed within 3 months prior to study entry must be greater or equal to 50% regardless of the facility's LLN.
* ECG performed within 4 weeks before study entry must demonstrate a QTc interval that is less than or equal to 0.47 seconds.
* The TSH level must be within normal limits for the laboratory.

Exclusion Criteria:

* Tumor that has been determined to be HER2-positive by immunohistochemistry (3+) or by FISH or CISH (positive for gene amplification), or has been determined to be HER2-equivocal and the investigator plans to administer trastuzumab or other targeted therapy.
* FNA alone to diagnose the primary breast cancer.
* Excisional biopsy or lumpectomy performed prior to study entry.
* Surgical axillary staging procedure prior to study entry.
* Definitive clinical or radiologic evidence of metastatic disease.
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral DCIS treated with RT.
* Contralateral invasive breast cancer at any time.
* Non-breast malignancies unless the patient is considered to be disease-free for 5 or more years prior to study entry and is deemed by her physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Requirement for chronic use of any of the prohibited medications or substances
* Previous therapy with anthracyclines, taxanes, or pazopanib for any malignancy.
* Treatment including RT, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to study entry.
* Continued therapy with any hormonal agent such as raloxifene, tamoxifen, or other SERM.
* Any sex hormonal therapy, e.g., birth control pills and ovarian hormone replacement therapy
* History of hepatitis B or C.
* Symptomatic pancreatitis or asymptomatic greater or equal to grade 2 elevation of amylase or lipase as per NCI CTCAE v3.0.
* History of documented pancreatitis.
* Uncontrolled hypertension defined as systolic BP greater than 140 mmHg or diastolic BP greater greater than 90 mmHg, with or without anti-hypertensive medication.
* History of hypertensive crisis or hypertensive encephalopathy.
* Cardiac disease that would preclude the use of any of the drugs included in the FB-6 treatment regimen.
* History of TIA or CVA.
* History of any arterial thrombotic event within 12 months prior to study entry.
* Pulmonary embolism or DVT within 6 months prior to study entry.
* Symptomatic peripheral vascular disease.
* Any significant bleeding within 6 months prior to study entry, exclusive of menorrhagia in premenopausal women.
* Known bleeding diathesis, coagulopathy, or requirement for therapeutic doses of coumadin.
* Serious or non-healing wound, skin ulcers, or bone fracture.
* Gastroduodenal ulcer(s) determined by endoscopy to be active.
* History of GI perforation, abdominal fistulae, or intra-abdominal abscess.
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal function.
* Sensory/motor neuropathy greater or equal to grade 2, as defined by the NCI's CTCAE v3.0.
* Conditions that would prohibit intermittent administration of corticosteroids for paclitaxel premedication.
* Anticipation of need for major surgical procedures (other than the required breast surgery) during the course of study therapy and for at least 3 months following the last dose of pazopanib.
* Pregnancy or lactation at the time of study entry.
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Known immediate or delayed hypersensitivity reaction to doxorubicin, cyclophosphamide, paclitaxel, pazopanib, or drugs chemically related to pazopanib.
* Use of any investigational agent within 4 weeks prior to enrollment in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (103):
- United States (100):
  - GSK Investigational Site, Decatur, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Richmond, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, San Rafael, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, South San Francisco, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Vacaville, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Greeley, Colorado
  - GSK Investigational Site, Lafayette, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Fernandina Beach, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orange Park, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Jeffersonville, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Battle Creek, Michigan
  - GSK Investigational Site, Brighton, Michigan
  - GSK Investigational Site, Byron Center, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Grosse Point Woods, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Livonia, Michigan
  - GSK Investigational Site, Mount Clemens, Michigan
  - GSK Investigational Site, Muskegon, Michigan
  - GSK Investigational Site, Port Huron, Michigan
  - GSK Investigational Site, Saginaw, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Warren, Michigan
  - GSK Investigational Site, Brunsville, Minnesota
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Maplewood, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Louis Park, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Clinton, North Carolina
  - GSK Investigational Site, Goldsboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Wilson, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Chargrin, Ohio
  - GSK Investigational Site, Clevand, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Lebanon, Ohio
  - GSK Investigational Site, Mentor, Ohio
  - GSK Investigational Site, Middletown, Ohio
  - GSK Investigational Site, Westlake, Ohio
  - GSK Investigational Site, Wilminton, Ohio
  - GSK Investigational Site, Xenia, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Ephrata, Pennsylvania
  - GSK Investigational Site, Greensburg, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, West Reading, Pennsylvania
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Vancover, Washington
  - GSK Investigational Site, Chippewa Falls, Wisconsin
  - GSK Investigational Site, Eau Claire, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin
  - GSK Investigational Site, Minocqua, Wisconsin
  - GSK Investigational Site, Rhinelander, Wisconsin
  - GSK Investigational Site, Rice Lake, Wisconsin
  - GSK Investigational Site, Stevens Point, Wisconsin
  - GSK Investigational Site, Weston, Wisconsin
  - GSK Investigational Site, Wisconsin Rapids, Wisconsin
- Canada (3):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib: Participants (par.) were treated with intravenous (IV) doxorubicin (60 milligrams per meters squared [mg/m^2]) and cyclophosphamide (AC) (600 mg/m^2) every 21 days for 4 cycles. This was followed by weekly paclitaxel (WP) 80 mg/m^2 IV on Days 1, 8, and 15 every 28 days for 4 cycles given concurrently with oral pazopanib 800 mg (2 tablets taken at the same time each day, either 1 hour before or 2 hours after a meal) taken daily and continuing until 7 days before surgery. Pazopanib was resumed at the same oral dose 4-6 weeks after surgery and was continued daily for 6 months.
Period: Doxorubicin and Cyclophosphamide (AC)
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Started | 101
Completed | 95
Not Completed | 6
Not completed — Disease Progression | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Participant Moved | 1
Period: Weekly Paclitaxel
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Started | 94 (One par. was deemed ineligible after completing AC therapy and did not start paclitaxel+pazopanib.)
Completed | 78
Not Completed | 16
Not completed — Disease Progression | 1
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Period: Pazopanib Presurgery Treatment (PPT)
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Started | 94
Completed | 36
Not Completed | 58
Not completed — Adverse Event | 52
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Never Started Pre-operative Pazopanib | 1
Period: Pazopanib Postsurgery Treatment
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Started | 42 (36 participants completed PPT; 7 participants who discontinued PPT resumed treatment postsurgery.)
Completed | 16
Not Completed | 26
Not completed — Adverse Event | 19
Not completed — Withdrawal by Subject | 5
Not completed — Moved | 1
Not completed — Site Thought Treatment Was Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib: Participants were treated with intravenous (IV) doxorubicin (60 milligrams per meters squared [mg/m^2]) and cyclophosphamide (AC) (600 mg/m^2) every 21 days for 4 cycles. This was followed by weekly paclitaxel (WP) 80 mg/m^2 IV on Days 1, 8, and 15 every 28 days for 4 cycles given concurrently with oral pazopanib 800 mg (2 tablets taken at the same time each day, either 1 hour before or 2 hours after a meal) taken daily and continuing until 7 days before surgery. Pazopanib was resumed at the same oral dose 4-6 weeks after surgery and was continued daily for 6 months.
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristic data are reported for members of the Treated Population, comprised of all participants who entered the study and received at least one dose of any study medication.
  Years | 50.9 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristic data are reported for members of the Treated Population, comprised of all participants who entered the study and received at least one dose of any study medication.
  Participants
    Female | 101
    Male | 0
Race/Ethnicity, Customized [Number; unit: participants] — Baseline Characteristic data are reported for members of the Treated Population, comprised of all participants who entered the study and received at least one dose of any study medication.
  participants
    White - White/Caucasian/European Heritage (W/C/EH) | 81
    African American/African Heritage | 10
    White - Arabic/North African Heritage | 3
    Asian - South East Asian Heritage | 3
    American Indian (AI) or Alaskan Native (AN) | 1
    Asian - Central/South Asian Heritage | 1
    Asian - East Asian Heritage | 1
    AI or AN + White - W/C/EH | 1
Number of participants with a positive or negative status for the indicated hormone receptors [Number; unit: participants] — Baseline Characteristic (BC) data are reported for members of the Treated Population. Receptor status is used to determine a course of treatment. Participants with hormone-receptor positive tumors could have been treated with hormonal therapy. Human epidermal growth factor receptor-2 (HER-2) is also known as NEU. Each participant was to be assessed for each tumor hormone receptor.
  participants
    Estrogen receptor (ER) status positive | 73
    ER status negative | 28
    Progesterone receptor (PgR) status positive | 62
    PgR status negative | 39
    HER-2/NEU status positive | 1
    HER-2/NEU status negative | 99
    HER-2/NEU status equivocal (uncertain) | 1
Number of participants with the indicted hormonal status (ER+ and PR+ / ER- and PR-) [Number; unit: participants] — BC data are reported for members of the Treated Population. Estrogen causes certain breast cancers (called ER+ cancers) to grow; these cancer cells have ERs on their surfaces. ER+ and PR+ indicate ER and PR positivity; a minus sign indicates that cells are negative for receptors. A participant's hormone status determines treatment modalities.
  participants
    Positive | 74
    Negative | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR) in the Breast and Nodes
Description: pCR was defined as no histologic evidence of invasive tumor cells in the surgical breast specimen, axillary nodes, or sentinel node identified after neoadjuvant chemotherapy.
Time Frame: From the start of the study until the time of surgery (average of 221.9 days [standard deviation of 23.65 days] after study entry)
Population: Evaluable Population: all participants who entered the study and received at least one dose of pazopanib.
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 93
Participants | 16
Statistical Analysis 1: Comparison: AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib; Test type: Superiority or Other; Percentage of participants = 17.98, 95% CI 2-sided [10.64 to 27.55] — The estimated value (EV) represents the percentage of participants with pCR. Participants with missing data were excluded from the denominator (n=89; 4 participants with missing data) for the calculation of the EV

2. Secondary Outcome: Number of Participants With Pathologic Complete Response (pCR) in the Breast
Description: pCR was defined as no histologic evidence of invasive tumor cells in the surgical breast specimen.
Time Frame: From the start of the study until the time of surgery (average of 221.9 [standard deviation of 23.65 days] days after study entry)
Population: Evaluable Population
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 93
Participants | 18

3. Secondary Outcome: Number of Participants With Clinical Complete Response (cCR) in the Breast and Nodes at the Completion of the Doxorubicin and Cyclophosphamide (AC) Period
Description: cCR was determined by tumor assessments performed by palpation. All clinical response assessments were to be performed by physical examination of the breast and the axilla. cCR was defined as the resolution of all target and non-target lesions identified at Baseline and no new lesions or other signs of disease progression. The criteria to be used for the determination of progressive disease were at the investigator's discretion.
Time Frame: From the start of the study until an average of 86.2 days (standard deviation of 5.76 days) after study entry
Population: Evaluable Population
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 93
Participants | 22

4. Secondary Outcome: Number of Participants With Clinical CR (cCR) in the Breast and Nodes at the Completion of the AC and Weekly Paclitaxel (WP) + Pazopanib Preoperative Periods
Description: as for outcome 3
Time Frame: From the start of the study until the preoperative evaluation (an average of 203.0 days [standard deviation of 23.19 days] after study entry)
Population: Evaluable Population
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 93
Participants | 39

5. Secondary Outcome: Invasive Recurrence-free Interval (IRFI)
Description: IRFI was assessed as the time from study entry until the diagnosis of the first invasive local (evidence of invasive/in situ breast cancer [except LCIS] in the ipsilateral breast [IB]/skin of the breast), regional (development of tumor in the ipsilateral [IP] internal mammary, IP supraclavicular, IP infraclavicular, and/or IP axillary nodes, as well as the soft tissue of the IP axilla, following surgery), or distant (evidence of tumor in all areas, with the exception of those described for local and regional recurrence) breast cancer recurrence during the 24 months after study entry.
Time Frame: up to 24 months after study entry
Population: Evaulable Population. Participants with recurrence before study entry were excluded from analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 92
months | NA [NA to NA] — The median was not estimable because too few participants had events.

6. Secondary Outcome: Number of Participants With Cardiac Toxicity (Per Common Terminology Criteria for Adverse Events Version 3) at the Completion of the AC Period
Description: The number of participants with cardiac toxicity was defined as those who had cardiac events of Grades (G) 3 and 4 leftventricular dysfunction (LVD) (CTCAE Version 3.0) and/or who had definite or probable cardiac death. Grade refers to the severity of the AE: G 1, mild AE; G 2, moderate AE; G 3, severe AE; G 4, life-threatening/disabling AE; G 5, death related to the AE. A G3 LVD event is defined as symptomatic congestive heart failure (CHF) responsive to intervention. A G4 event is defined as poorly controlled refractory CHF; ventricular assist device or heart transplant indicated.
Time Frame: From the start of the study until the preoperative evaluation (an average of 86.2 days [standard deviation of 5.76 days] after study entry)
Population: Treated Population: all participants who entered the study and received at least one dose of any study medication
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 101
Participants | 0

7. Secondary Outcome: Number of Participants With Cardiac Toxicity (Per CTCAE Version 3) at the Completion of the AC and Weekly Paclitaxel (WP) + Pazopanib Preoperative Periods
Description: as for outcome 6
Time Frame: as for outcome 4
Population: Treated Population
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 101
Participants | 0

8. Secondary Outcome: Number of Participants With Cardiac Toxicity (Per CTCAE Version 3.0) During the Postoperative Pazopanib Period
Description: as for outcome 6
Time Frame: From the start of the study until the end of the postoperative pazopanib period, which coincides with the start of the end of treatment period (an average of 310.8 days [standard deviation of 85.29 days] after study entry)
Population: Treated Population: Only those members of the Treated Population who started the postoperative pazopanib period were assessed.
Measure: Number; unit: Participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 42
Participants | 0

9. Secondary Outcome: Participants With Normal Thyroid Stimulating Hormone (TSH) Levels at Baseline Who Had an Elevated TSH Level at Least Once During the Study and During the Individual Study Periods
Description: The number of participants with normal thyroid function at Baseline who had an elevation in TSH during the study were recorded. TSH elevation was derived based on local laboratory ranges.
Time Frame: up to 24 months after study entry
Population: Treated Population. Data are presented for only those participants who remained in the study during the indicated period and had their blood drawn for assessment.
Measure: Number; unit: participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 101
participants
  Elevated TSH at Least Once during the Study, n=101 | 28
  AC Period, n=91 | 2
  (WP) + Pazopanib Preoperative Periods, n=89 | 15
  Surgery Period, n=78 | 1
  Postoperative Pazopanib Period, n=36 | 7
  Follow-up Period, n=33 | 8

10. Secondary Outcome: Number of Participants With the Indicated Radiotherapy-related Complications
Time Frame: up to 24 months after study entry
Population: Treated Population
Measure: Number; unit: participants
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 101
participants
  Rash | 57
  Pneumonitis | 1

11. Secondary Outcome: Number of Participants With Recurrence Events
Description: The number of participants with recurrence events during the 24 months after study entry are reported. A recurrence event is defined as invasive local (evidence of invasive/in situ breast cancer [except LCIS] in the ipsilateral breast [IB]/skin of the breast), regional (development of tumor in the ipsilateral [IP] internal mammary, IP supraclavicular, IP infraclavicular, and/or IP axillary nodes, as well as the soft tissue of the IP axilla, following surgery), or distant (evidence of tumor in all areas, with the exception of those described for local and regional recurrence) breast cancer recurrence during the 24 months after study entry.
Time Frame: up to 24 months after study entry
Population: Evaulable Population, excluding participants with recurrence before study entry
Measure: Number; unit: participants
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Number analyzed (Participants) | 92
participants | 15

ADVERSE EVENTS:
Arm/Group | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib
Serious Adverse Events (participants affected / at risk) | 15/101
Other Adverse Events (participants affected / at risk) | 101/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib (N=101)
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Perineal abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Convulsion (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AC, Followed by Weekly Paclitaxel and Concurrent Pazopanib (N=101)
Nausea (Gastrointestinal disorders) | 72
Diarrhoea (Gastrointestinal disorders) | 69
Constipation (Gastrointestinal disorders) | 55
Vomiting (Gastrointestinal disorders) | 34
Stomatitis (Gastrointestinal disorders) | 25
Dyspepsia (Gastrointestinal disorders) | 22
Oral pain (Gastrointestinal disorders) | 13
Flatulence (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 10
Haemorrhoids (Gastrointestinal disorders) | 7
Toothache (Gastrointestinal disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 93
Pain (Gastrointestinal disorders) | 30
Pyrexia (General disorders) | 19
Mucosal inflammation (General disorders) | 18
Oedema peripheral (General disorders) | 8
Influenza like illness (General disorders) | 7
Chills (General disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 70
Nail disorder (Skin and subcutaneous tissue disorders) | 19
Rash (Skin and subcutaneous tissue disorders) | 17
Erythema (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 13
Dry skin (Skin and subcutaneous tissue disorders) | 7
Nail discolouration (Skin and subcutaneous tissue disorders) | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 45
Headache (Nervous system disorders) | 36
Neuropathy peripheral (Nervous system disorders) | 22
Paraesthesia (Nervous system disorders) | 21
Dizziness (Nervous system disorders) | 20
Peripheral sensory neuropathy (Nervous system disorders) | 18
Hypoaesthesia (Nervous system disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24
Neutrophil count decreased (Investigations) | 37
Alanine aminotransferase increased (Investigations) | 15
Weight decreased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 13
Weight increased (Investigations) | 8
White blood cell count decreased (Investigations) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Back pain (Musculoskeletal and connective tissue disorders) | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Hot flush (Vascular disorders) | 40
Hypertension (Vascular disorders) | 30
Infection (Infections and infestations) | 17
Nasopharyngitis (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 6
Insomnia (Psychiatric disorders) | 33
Anxiety (Psychiatric disorders) | 17
Depression (Psychiatric disorders) | 9
Mood altered (Psychiatric disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 31
Dehydration (Metabolism and nutrition disorders) | 7
Radiation skin injury (Injury, poisoning and procedural complications) | 10
Seroma (Injury, poisoning and procedural complications) | 10
Vision blurred (Eye disorders) | 11
Lacrimation increased (Eye disorders) | 7
Breast pain (Reproductive system and breast disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 13
Hypothyroidism (Endocrine disorders) | 12
Ear pain (Ear and labyrinth disorders) | 9
Palpitations (Cardiac disorders) | 8
Dysuria (Renal and urinary disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.